CLINICAL TRIAL: NCT03912883
Title: Prognostic Factors in Prostate Cancer for Patients Treated by Watchful Waiting
Acronym: TAPG
Status: Active, not recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 005937
Record Dates: First submitted 2019-02-14; First posted 2019-04-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: biomarkers; pathology; tissue; watchful waiting; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — H&E slides and/or FFPE blocks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Trans-Atlantic Prostate Group (TAPG) was established to examine the hypothesis that through a detailed retrospective analysis of outcome in a group of men with clinically localised prostate cancer at diagnosis, variables such as biological, pathological and clinical markers, could be identified that might accurately predict the prognosis of clinically localised prostate cancer.

DETAILED DESCRIPTION:
In 1999, the TAPG group initiated the "Prognostic Factors in Prostate Cancer for Patients Treated by Watchful Waiting" study, referred to as the TAPG study. It is a retrospective population-based tissue sample study in men diagnosed with localised prostate cancer 1990-2006, inclusively. Initially the cohort comprised men diagnosed with prostate cancer with transurethral resection of the prostate (TURP) and needle biopsies 1990-1996, but was expanded from 2005 to include men diagnosed with prostate cancer 1990 - 2006. Data was collected from six regional cancer registries and eligibility was confirmed via hospital sites, which sent the relevant tissue samples to the TAPG Central Coordinating Office (CCO). Selection of eligible patients for the study completed in 2010. Since this year the TAPG CCO has been collecting cancer registration and mortality updates on the cohort members from regional cancer registries.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged less than 76 years at the time of diagnosis
* Patients must have had a baseline serum PSA level measured before starting any treatment and within six months of diagnosis
* Patients must have been diagnosed between 1990 and 2006 with a clinically localized (clinical stage T1-T3, N0 or NX, MO or MX) prostate cancer, in the judgment of the treating physician
* The initial diagnostic biopsy sample must be available for review. Patients should have (but are not required to have) tissue blocks available for review.
* There must be no evidence of metastatic disease
* While data collection will include review of the reports of any imaging studies of the prostate, bones, or soft tissues, these studies are not essential
* Each patient should have had an adequate medical evaluation to document the status of disease for the first five years after diagnosis. Follow-up should include an annual PSA and digital rectal examination. Records will be reviewed to seek all information about medical evaluation after the time of diagnosis.

Exclusion Criteria:

* Patients older than 76 years at the time of diagnosis
* Patients who have not had a baseline serum PSA level measured before starting any treatment
* Patients who do not have the initial diagnosis biopsy sample for review
* Patients with evidence of metastatic disease

Ages: 18 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective, exploratory cohort study and will be carried out in patients registered on UK regional cancer registry databases, as having been diagnosed with prostate cancer between 1990 and 2006, inclusive.
Sampling Method: Non-Probability Sample
Enrollment: 3350 (Estimated)
Dates: Start 1999-10-12 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-specific survival | From date of inclusion to date of death from prostate cancer, assessed up to 30 years.
  Time from date of inclusion until death from prostate cancer.
Overall survival | From date of inclusion to date of death from any cause, assessed up to 30 years.
  Time from date of inclusion until death from any cause.

SECONDARY OUTCOMES:
To evaluate a correlation between serum PSA level and prostate cancer-specific survival. | From date of inclusion to date of death from prostate cancer, assessed up to 30 years.
  Correlation of serum PSA level taken within 6 months of date of inclusion compared to death from prostate cancer.
To evaluate a correlation between Gleason score and prostate cancer-specific survival. | From date of inclusion to date of death from prostate cancer, assessed up to 30 years.
  Correlation of Gleason Score at date of inclusion compared to death from prostate cancer.
To evaluate an association between clinical stage and prostate cancer-specific survival. | From date of inclusion to date of death from any cause, assessed up to 30 years.
  Stratification of clinical stage at date of inclusion compared to death from prostate cancer.
To evaluate ki-67-positive biomarker predictors of prognosis in early prostate cancer. | From date of inclusion to date of death from prostate cancer, assessed up to 30 years.
  Correlation of ki-67-positive cells compared to prostate cancer-specific survival.
To evaluate ki-67-positive biomarker predictors of prognosis in early prostate cancer. | From date of inclusion to date of death from any cause, assessed up to 30 years.
  Correlation of ki-67-positive cells compared to overall cancer-specific survival.
To evaluate ERG-ETV1 biomarker predictors of prognosis in early prostate cancer. | From date of inclusion to date of death from prostate cancer, assessed up to 30 years.
  Correlation of ERG-ETV1 rearrangement status compared to prostate cancer-specific survival.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beltran L, Ahmad AS, Sandu H, Kudahetti S, Soosay G, Moller H, Cuzick J, Berney DM; Transatlantic Prostate Group. Histopathologic False-positive Diagnoses of Prostate Cancer in the Age of Immunohistochemistry. Am J Surg Pathol. 2019 Mar;43(3):361-368. doi: 10.1097/PAS.0000000000001202. PMID 30531531
- [Background] Ahmad AS, Parameshwaran V, Beltran L, Fisher G, North BV, Greenberg D, Soosay G, Moller H, Scardino P, Cuzick J, Berney DM; Transatlantic Prostate Group. Should reporting of peri-neural invasion and extra prostatic extension be mandatory in prostate cancer biopsies? correlation with outcome in biopsy cases treated conservatively. Oncotarget. 2018 Apr 17;9(29):20555-20562. doi: 10.18632/oncotarget.24994. eCollection 2018 Apr 17. PMID 29755671
- [Background] Stankiewicz E, Mao X, Mangham DC, Xu L, Yeste-Velasco M, Fisher G, North B, Chaplin T, Young B, Wang Y, Kaur Bansal J, Kudahetti S, Spencer L, Foster CS, Moller H, Scardino P, Oliver RT, Shamash J, Cuzick J, Cooper CS, Berney DM, Lu YJ. Identification of FBXL4 as a Metastasis Associated Gene in Prostate Cancer. Sci Rep. 2017 Jul 11;7(1):5124. doi: 10.1038/s41598-017-05209-z. PMID 28698647
- [Background] Berney DM, Beltran L, Fisher G, North BV, Greenberg D, Moller H, Soosay G, Scardino P, Cuzick J. Validation of a contemporary prostate cancer grading system using prostate cancer death as outcome. Br J Cancer. 2016 May 10;114(10):1078-83. doi: 10.1038/bjc.2016.86. Epub 2016 Apr 21. PMID 27100731
- [Background] Ahmad AS, Vasiljevic N, Carter P, Berney DM, Moller H, Foster CS, Cuzick J, Lorincz AT. A novel DNA methylation score accurately predicts death from prostate cancer in men with low to intermediate clinical risk factors. Oncotarget. 2016 Nov 1;7(44):71833-71840. doi: 10.18632/oncotarget.12377. PMID 27708246
- [Background] Cuzick J, Stone S, Fisher G, Yang ZH, North BV, Berney DM, Beltran L, Greenberg D, Moller H, Reid JE, Gutin A, Lanchbury JS, Brawer M, Scardino P. Validation of an RNA cell cycle progression score for predicting death from prostate cancer in a conservatively managed needle biopsy cohort. Br J Cancer. 2015 Jul 28;113(3):382-9. doi: 10.1038/bjc.2015.223. Epub 2015 Jun 23. PMID 26103570
- [Background] Vasiljevic N, Ahmad AS, Thorat MA, Fisher G, Berney DM, Moller H, Foster CS, Cuzick J, Lorincz AT. DNA methylation gene-based models indicating independent poor outcome in prostate cancer. BMC Cancer. 2014 Sep 6;14:655. doi: 10.1186/1471-2407-14-655. PMID 25193387
- [Background] Vasiljevic N, Ahmad AS, Carter PD, Fisher G, Berney DM, Foster CS, Cuzick J, Lorincz AT. DNA methylation of PITX2 predicts poor survival in men with prostate cancer. Biomark Med. 2014;8(9):1143-50. doi: 10.2217/bmm.14.41. PMID 25402584
- [Background] Merson S, Yang ZH, Brewer D, Olmos D, Eichholz A, McCarthy F, Fisher G, Kovacs G, Berney DM, Foster CS, Moller H, Scardino P, Cuzick J, Cooper CS, Clark JP; Transatlantic Prostate Group. Focal amplification of the androgen receptor gene in hormone-naive human prostate cancer. Br J Cancer. 2014 Mar 18;110(6):1655-62. doi: 10.1038/bjc.2014.13. Epub 2014 Jan 30. PMID 24481405
- [Background] Vasiljevic N, Ahmad AS, Beesley C, Thorat MA, Fisher G, Berney DM, Moller H, Yu Y, Lu YJ, Cuzick J, Foster CS, Lorincz AT. Association between DNA methylation of HSPB1 and death in low Gleason score prostate cancer. Prostate Cancer Prostatic Dis. 2013 Mar;16(1):35-40. doi: 10.1038/pcan.2012.47. Epub 2012 Nov 20. PMID 23165430
- [Background] Fisher G, Yang ZH, Kudahetti S, Moller H, Scardino P, Cuzick J, Berney DM; Transatlantic Prostate Group. Prognostic value of Ki-67 for prostate cancer death in a conservatively managed cohort. Br J Cancer. 2013 Feb 5;108(2):271-7. doi: 10.1038/bjc.2012.598. Epub 2013 Jan 17. PMID 23329234
- [Background] Cuzick J, Yang ZH, Fisher G, Tikishvili E, Stone S, Lanchbury JS, Camacho N, Merson S, Brewer D, Cooper CS, Clark J, Berney DM, Moller H, Scardino P, Sangale Z; Transatlantic Prostate Group. Prognostic value of PTEN loss in men with conservatively managed localised prostate cancer. Br J Cancer. 2013 Jun 25;108(12):2582-9. doi: 10.1038/bjc.2013.248. Epub 2013 May 21. PMID 23695019
- [Background] Ahmad I, Singh LB, Yang ZH, Kalna G, Fleming J, Fisher G, Cooper C, Cuzick J, Berney DM, Moller H, Scardino P, Leung HY. Mir143 expression inversely correlates with nuclear ERK5 immunoreactivity in clinical prostate cancer. Br J Cancer. 2013 Jan 15;108(1):149-54. doi: 10.1038/bjc.2012.510. PMID 23321517
- [Background] Jeetle SS, Fisher G, Yang ZH, Stankiewicz E, Moller H, Cooper CS, Cuzick J, Berney DM; Trans-Atlantic Prostate Group. Neuroendocrine differentiation does not have independent prognostic value in conservatively treated prostate cancer. Virchows Arch. 2012 Aug;461(2):103-7. doi: 10.1007/s00428-012-1259-2. Epub 2012 Jul 6. PMID 22767265
- [Background] Cuzick J, Berney DM, Fisher G, Mesher D, Moller H, Reid JE, Perry M, Park J, Younus A, Gutin A, Foster CS, Scardino P, Lanchbury JS, Stone S; Transatlantic Prostate Group. Prognostic value of a cell cycle progression signature for prostate cancer death in a conservatively managed needle biopsy cohort. Br J Cancer. 2012 Mar 13;106(6):1095-9. doi: 10.1038/bjc.2012.39. Epub 2012 Feb 23. PMID 22361632
- [Background] Rajab R, Fisher G, Kattan MW, Foster CS, Moller H, Oliver T, Reuter V, Scardino PT, Cuzick J, Berney DM; Transatlantic Prostate Group. An improved prognostic model for stage T1a and T1b prostate cancer by assessments of cancer extent. Mod Pathol. 2011 Jan;24(1):58-63. doi: 10.1038/modpathol.2010.182. Epub 2010 Sep 10. PMID 20834240
- [Background] O'Brien MF, Cronin AM, Fearn PA, Savage CJ, Smith B, Stasi J, Scardino PT, Fisher G, Cuzick J, Moller H, Oliver RT, Berney DM, Foster CS, Eastham JA, Vickers AJ, Lilja H; Trans-Atlantic Prostate Group. Evaluation of prediagnostic prostate-specific antigen dynamics as predictors of death from prostate cancer in patients treated conservatively. Int J Cancer. 2011 May 15;128(10):2373-81. doi: 10.1002/ijc.25570. PMID 20658531
- [Background] Cuzick J, Swanson GP, Fisher G, Brothman AR, Berney DM, Reid JE, Mesher D, Speights VO, Stankiewicz E, Foster CS, Moller H, Scardino P, Warren JD, Park J, Younus A, Flake DD 2nd, Wagner S, Gutin A, Lanchbury JS, Stone S; Transatlantic Prostate Group. Prognostic value of an RNA expression signature derived from cell cycle proliferation genes in patients with prostate cancer: a retrospective study. Lancet Oncol. 2011 Mar;12(3):245-55. doi: 10.1016/S1470-2045(10)70295-3. PMID 21310658
- [Background] Yao S, Bee A, Brewer D, Dodson A, Beesley C, Ke Y, Ambroisine L, Fisher G, Moller H, Dickinson T, Gerard P, Lian LY, Risk J, Lane B, Smith P, Reuter V, Berney D, Gosden C, Scardino P, Cuzick J, Djamgoz MB, Cooper C, Foster CS. PRKC-zeta Expression Promotes the Aggressive Phenotype of Human Prostate Cancer Cells and Is a Novel Target for Therapeutic Intervention. Genes Cancer. 2010 May;1(5):444-64. doi: 10.1177/1947601910376079. PMID 21779455
- [Background] Thomsen MK, Ambroisine L, Wynn S, Cheah KS, Foster CS, Fisher G, Berney DM, Moller H, Reuter VE, Scardino P, Cuzick J, Ragavan N, Singh PB, Martin FL, Butler CM, Cooper CS, Swain A; Transatlantic Prostate Group. SOX9 elevation in the prostate promotes proliferation and cooperates with PTEN loss to drive tumor formation. Cancer Res. 2010 Feb 1;70(3):979-87. doi: 10.1158/0008-5472.CAN-09-2370. Epub 2010 Jan 26. PMID 20103652
- [Background] Shan L, Ambroisine L, Clark J, Yanez-Munoz RJ, Fisher G, Kudahetti SC, Yang J, Kia S, Mao X, Fletcher A, Flohr P, Edwards S, Attard G, De-Bono J, Young BD, Foster CS, Reuter V, Moller H, Oliver TD, Berney DM, Scardino P, Cuzick J, Cooper CS, Lu YJ; Transatlantic Prostate Group. The identification of chromosomal translocation, t(4;6)(q22;q15), in prostate cancer. Prostate Cancer Prostatic Dis. 2010 Jun;13(2):117-25. doi: 10.1038/pcan.2010.2. Epub 2010 Feb 23. PMID 20177423
- [Background] Reid AH, Attard G, Ambroisine L, Fisher G, Kovacs G, Brewer D, Clark J, Flohr P, Edwards S, Berney DM, Foster CS, Fletcher A, Gerald WL, Moller H, Reuter VE, Scardino PT, Cuzick J, de Bono JS, Cooper CS; Transatlantic Prostate Group. Molecular characterisation of ERG, ETV1 and PTEN gene loci identifies patients at low and high risk of death from prostate cancer. Br J Cancer. 2010 Feb 16;102(4):678-84. doi: 10.1038/sj.bjc.6605554. Epub 2010 Jan 26. PMID 20104229
- [Background] Rajab R, Fisher G, Kattan MW, Foster CS, Oliver T, Moller H, Reuter V, Scardino P, Cuzick J, Berney DM; Transatlantic Prostate Group. Measurements of cancer extent in a conservatively treated prostate cancer biopsy cohort. Virchows Arch. 2010 Nov;457(5):547-53. doi: 10.1007/s00428-010-0971-z. Epub 2010 Sep 9. PMID 20827488
- [Background] Kudahetti SC, Fisher G, Ambroisine L, Prowse D, Kattan MW, Foster CS, Moller H, Oliver T, Fletcher A, Cooper C, Reuter V, Scardino P, Cuzick J, Berney DM; Transatlantic Prostate Group. Immunohistochemistry for p16, but not Rb or p21, is an independent predictor of prognosis in conservatively treated, clinically localised prostate cancer. Pathology. 2010;42(6):519-23. doi: 10.3109/00313025.2010.508788. PMID 20854069
- [Background] Kudahetti S, Fisher G, Ambroisine L, Foster C, Reuter V, Eastham J, Moller H, Kattan MW, Cooper CS, Scardino P, Cuzick J, Berney DM. p53 immunochemistry is an independent prognostic marker for outcome in conservatively treated prostate cancer. BJU Int. 2009 Jul;104(1):20-4. doi: 10.1111/j.1464-410X.2009.08407.x. Epub 2009 Feb 23. PMID 19239456
- [Background] Foster CS, Dodson AR, Ambroisine L, Fisher G, Moller H, Clark J, Attard G, De-Bono J, Scardino P, Reuter VE, Cooper CS, Berney DM, Cuzick J. Hsp-27 expression at diagnosis predicts poor clinical outcome in prostate cancer independent of ETS-gene rearrangement. Br J Cancer. 2009 Oct 6;101(7):1137-44. doi: 10.1038/sj.bjc.6605227. Epub 2009 Aug 25. PMID 19707199
- [Background] Berney DM, Gopalan A, Kudahetti S, Fisher G, Ambroisine L, Foster CS, Reuter V, Eastham J, Moller H, Kattan MW, Gerald W, Cooper C, Scardino P, Cuzick J. Ki-67 and outcome in clinically localised prostate cancer: analysis of conservatively treated prostate cancer patients from the Trans-Atlantic Prostate Group study. Br J Cancer. 2009 Mar 24;100(6):888-93. doi: 10.1038/sj.bjc.6604951. PMID 19293807
- [Background] Kattan MW, Cuzick J, Fisher G, Berney DM, Oliver T, Foster CS, Moller H, Reuter V, Fearn P, Eastham J, Scardino PT; Transatlantic Prostate Group. Nomogram incorporating PSA level to predict cancer-specific survival for men with clinically localized prostate cancer managed without curative intent. Cancer. 2008 Jan 1;112(1):69-74. doi: 10.1002/cncr.23106. PMID 18000803
- [Background] Eastham JA, Kattan MW, Fearn P, Fisher G, Berney DM, Oliver T, Foster CS, Moller H, Reuter V, Cuzick J, Scardino P; Transatlantic Prostate Group. Local progression among men with conservatively treated localized prostate cancer: results from the Transatlantic Prostate Group. Eur Urol. 2008 Feb;53(2):347-54. doi: 10.1016/j.eururo.2007.05.015. Epub 2007 May 30. PMID 17544572
- [Background] Clark J, Attard G, Jhavar S, Flohr P, Reid A, De-Bono J, Eeles R, Scardino P, Cuzick J, Fisher G, Parker MD, Foster CS, Berney D, Kovacs G, Cooper CS. Complex patterns of ETS gene alteration arise during cancer development in the human prostate. Oncogene. 2008 Mar 27;27(14):1993-2003. doi: 10.1038/sj.onc.1210843. Epub 2007 Oct 8. PMID 17922029
- [Background] Attard G, Clark J, Ambroisine L, Mills IG, Fisher G, Flohr P, Reid A, Edwards S, Kovacs G, Berney D, Foster C, Massie CE, Fletcher A, De Bono JS, Scardino P, Cuzick J, Cooper CS; Transatlantic Prostate Group. Heterogeneity and clinical significance of ETV1 translocations in human prostate cancer. Br J Cancer. 2008 Jul 22;99(2):314-20. doi: 10.1038/sj.bjc.6604472. Epub 2008 Jul 1. PMID 18594527
- [Background] Attard G, Clark J, Ambroisine L, Fisher G, Kovacs G, Flohr P, Berney D, Foster CS, Fletcher A, Gerald WL, Moller H, Reuter V, De Bono JS, Scardino P, Cuzick J, Cooper CS; Transatlantic Prostate Group. Duplication of the fusion of TMPRSS2 to ERG sequences identifies fatal human prostate cancer. Oncogene. 2008 Jan 10;27(3):253-63. doi: 10.1038/sj.onc.1210640. Epub 2007 Jul 16. PMID 17637754
- [Background] Berney DM, Fisher G, Kattan MW, Oliver RT, Moller H, Fearn P, Eastham J, Scardino P, Cuzick J, Reuter VE, Foster CS; Trans-Atlantic Prostate Group. Major shifts in the treatment and prognosis of prostate cancer due to changes in pathological diagnosis and grading. BJU Int. 2007 Dec;100(6):1240-4. doi: 10.1111/j.1464-410X.2007.07199.x. PMID 17979924
- [Background] Berney DM, Fisher G, Kattan MW, Oliver RT, Moller H, Fearn P, Eastham J, Scardino P, Cuzick J, Reuter VE, Foster CS; Trans-Atlantic prostate group. Pitfalls in the diagnosis of prostatic cancer: retrospective review of 1791 cases with clinical outcome. Histopathology. 2007 Oct;51(4):452-7. doi: 10.1111/j.1365-2559.2007.02819.x. PMID 17880526
- [Background] Cuzick J, Fisher G, Kattan MW, Berney D, Oliver T, Foster CS, Moller H, Reuter V, Fearn P, Eastham J, Scardino P; Transatlantic Prostate Group. Long-term outcome among men with conservatively treated localised prostate cancer. Br J Cancer. 2006 Nov 6;95(9):1186-94. doi: 10.1038/sj.bjc.6603411. PMID 17077805
- [Background] Kammerer-Jacquet SF, Ahmad A, Moller H, Sandu H, Scardino P, Soosay G, Beltran L, Cuzick J, Berney DM. Ki-67 is an independent predictor of prostate cancer death in routine needle biopsy samples: proving utility for routine assessments. Mod Pathol. 2019 Sep;32(9):1303-1309. doi: 10.1038/s41379-019-0268-y. Epub 2019 Apr 11. PMID 30976102
- [Background] Berney DM, Beltran L, Sandu H, Soosay G, Moller H, Scardino P, Murphy J, Ahmad A, Cuzick J; Transatlantic Prostate Group. The percentage of high-grade prostatic adenocarcinoma in prostate biopsies significantly improves on Grade Groups in the prediction of prostate cancer death. Histopathology. 2019 Oct;75(4):589-597. doi: 10.1111/his.13888. Epub 2019 Aug 13. PMID 31032963